CLINICAL TRIAL: NCT01751789
Title: Linking Opioid Dependent Patients From Inpatient Detoxification to Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA034261
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Illicit Opioid Drug Use
Keywords: illicit opioid drug use; health service utilization
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Genetic Linkage; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linkage (Active Comparator): Participants will receive Suboxone during their inpatient detoxication and be given outpatient appointments to continue Suboxone treatment after completing inpatient detoxification
  Interventions: Behavioral: Linkage
- Detoxification (Placebo Comparator): Participants will receive Suboxone to detoxify from opioids and the standard treatment offered by the inpatient detoxification program
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Linkage
  Arms: Linkage
Other: Treatment as Usual
  Arms: Detoxification

SUMMARY:
The purpose of this study is to determine whether, for individuals in inpatient opioid detoxification, linking to outpatient Suboxone treatment increases treatment adherence and reduces relapse to illicit opioid use.

DETAILED DESCRIPTION:
In this randomized trial, consenting individuals seeking inpatient opioid detoxification will be assigned to one of two groups. The first group will receive a tapering schedule of buprenorphine during inpatient detoxification to alleviate acute withdrawal symptoms, and referral to a community medical and substance abuse treatment providers (DETOX). The second group will also receive buprenorphine to relieve withdrawal symptoms, but will maintain a stable dose of buprenorphine through inpatient discharge and linkage to an appointment with a primary care provider within a week of discharge (LINKAGE). All participants complete study assessments at baseline, 1-month, 3-months and 6-months post-enrollment.

The SSTAR inpatient detoxification program based in Fall River, Massachusetts will serve as the recruitment site of this trial. SSTAR's program has 38 beds and is a 24-hour medically and psychiatrically supervised treatment facility that provides evaluation and withdrawal management. The SSTAR Family Healthcare Center is a 330 Federally Qualified facility also in Fall River that provides primary care and behavioral health services to residents of Community Health Network Area 25 (Fall River, Somerset, Swansea and Westport, Massachusetts). Dr. Bailey, Director of Research at SSTAR, will oversee the provision of buprenorphine treatment to study participants during detoxification and serve as liaison to the primary care providers at the Family Healthcare Center.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* opioid dependent;
* interested in initiating maintenance buprenorphine treatment;
* opioid positive on urine toxicology;
* willing to establish primary care with a buprenorphine-waivered physician at SSTAR.

Exclusion Criteria:

* Patients unable to provide informed consent due to acute illness, cognitive impairment, or psychosis;
* probation/parole requirements that might interfere with protocol participation (1% of SSTAR inpatients);
* inability to provide two contact persons to verify location;
* not able to complete assessments in English;
* currently enrolled in a methadone or suboxone maintenance program;
* plans to leave the area within the next 6 months;
* current DSM-IV diagnosis of substance dependence for sedative/hypnotic drugs, cocaine, or alcohol;
* current suicidality on the Modified Scale for Suicidal Ideation;
* chronic pain requiring ongoing opioid use or anticipated major painful event (significant surgical procedure) in the coming 6 months;
* pregnancy;
* history of allergic reaction to buprenorphine or naloxone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Illicit opioid use | 6 months
  Illicit opioid use will be measured by self-report and by urine toxicology
Health Service Utilization | 6 months
  Health service utilization will be measured by self-report and medical chart review

CONTACTS AND LOCATIONS:
Locations (1):
- SSTAR, Fall River, Massachusetts, United States

REFERENCES:
- [Derived] Christopher PP, Anderson B, Stein MD. Comparing views on civil commitment for drug misuse and for mental illness among persons with opioid use disorder. J Subst Abuse Treat. 2020 Jun;113:107998. doi: 10.1016/j.jsat.2020.107998. Epub 2020 Mar 5. PMID 32359671
- [Derived] Stein MD, Kenney SR, Anderson BJ, Conti MT, Bailey GL. Prescribed and non-prescribed gabapentin use among persons seeking inpatient opioid detoxification. J Subst Abuse Treat. 2020 Mar;110:37-41. doi: 10.1016/j.jsat.2019.12.007. Epub 2019 Dec 13. PMID 31952626
- [Derived] Stein MD, Kenney SR, Anderson BJ, Bailey GL. Perceptions about fentanyl-adulterated heroin and overdose risk reduction behaviors among persons seeking treatment for heroin use. J Subst Abuse Treat. 2019 Sep;104:144-147. doi: 10.1016/j.jsat.2019.07.006. Epub 2019 Jul 13. PMID 31370978
- [Derived] Pivovarova E, Stein MD. In their own words: language preferences of individuals who use heroin. Addiction. 2019 Oct;114(10):1785-1790. doi: 10.1111/add.14699. Epub 2019 Jul 11. PMID 31140667
- [Derived] Kenney SR, Anderson BJ, Bailey GL, Stein MD. Drug Use-Related Normative Misperceptions and Behaviors Among Persons Seeking Heroin Withdrawal Management. J Addict Med. 2019 May/Jun;13(3):215-219. doi: 10.1097/ADM.0000000000000482. PMID 30461441
- [Derived] Christopher PP, Anderson B, Stein MD. Civil commitment experiences among opioid users. Drug Alcohol Depend. 2018 Dec 1;193:137-141. doi: 10.1016/j.drugalcdep.2018.10.001. Epub 2018 Oct 18. PMID 30384320
- [Derived] Kenney SR, Anderson BJ, Bailey GL, Stein MD. Buprenorphine treatment formulations: Preferences among persons in opioid withdrawal management. J Subst Abuse Treat. 2018 Nov;94:55-59. doi: 10.1016/j.jsat.2018.08.011. Epub 2018 Aug 28. PMID 30243418
- [Derived] Stein MD, Kenney SR, Anderson BJ, Bailey GL. Loaded: Gun involvement among opioid users. Drug Alcohol Depend. 2018 Jun 1;187:205-211. doi: 10.1016/j.drugalcdep.2018.03.015. Epub 2018 Apr 16. PMID 29680676
- [Derived] Kenney SR, Anderson BJ, Conti MT, Bailey GL, Stein MD. Expected and actual fentanyl exposure among persons seeking opioid withdrawal management. J Subst Abuse Treat. 2018 Mar;86:65-69. doi: 10.1016/j.jsat.2018.01.005. Epub 2018 Jan 4. PMID 29415853
- [Derived] Kenney SR, Anderson BJ, Stein MD. Drinking to cope mediates the relationship between depression and alcohol risk: Different pathways for college and non-college young adults. Addict Behav. 2018 May;80:116-123. doi: 10.1016/j.addbeh.2018.01.023. Epub 2018 Feb 4. PMID 29407681
- [Derived] Stein MD, Conti MT, Kenney S, Anderson BJ, Flori JN, Risi MM, Bailey GL. Adverse childhood experience effects on opioid use initiation, injection drug use, and overdose among persons with opioid use disorder. Drug Alcohol Depend. 2017 Oct 1;179:325-329. doi: 10.1016/j.drugalcdep.2017.07.007. Epub 2017 Aug 5. PMID 28841495
- [Derived] Stein MD, Flori JN, Risi MM, Conti MT, Anderson BJ, Bailey GL. Overdose history is associated with postdetoxification treatment preference for persons with opioid use disorder. Subst Abus. 2017 Oct-Dec;38(4):389-393. doi: 10.1080/08897077.2017.1353570. Epub 2017 Jul 10. PMID 28692407
- [Derived] Kenney SR, Anderson BJ, Bailey GL, Stein MD. The relationship between diversion-related attitudes and sharing and selling buprenorphine. J Subst Abuse Treat. 2017 Jul;78:43-47. doi: 10.1016/j.jsat.2017.04.017. Epub 2017 Apr 27. PMID 28554602
- [Derived] Kenney SR, Bailey GL, Anderson BJ, Stein MD. Heroin refusal self-efficacy and preference for medication-assisted treatment after inpatient detoxification. Addict Behav. 2017 Oct;73:124-128. doi: 10.1016/j.addbeh.2017.05.009. Epub 2017 May 9. PMID 28505487
- [Derived] Stein MD, Anderson BJ, Kenney SR, Bailey GL. Beliefs about the consequences of using benzodiazepines among persons with opioid use disorder. J Subst Abuse Treat. 2017 Jun;77:67-71. doi: 10.1016/j.jsat.2017.03.002. Epub 2017 Mar 9. PMID 28476275
- [Derived] Schonbrun YC, Anderson BJ, Johnson JE, Stein MD. Feasibility of a Supportive Other Intervention for Opiate-Dependent Patients Entering Inpatient Detoxification. J Psychoactive Drugs. 2016 Jul-Aug;48(3):181-6. doi: 10.1080/02791072.2016.1179377. Epub 2016 May 16. PMID 27182836
- [Derived] Stein MD, Anderson BJ, Bailey GL. Preferences for Aftercare Among Persons Seeking Short-Term Opioid Detoxification. J Subst Abuse Treat. 2015 Dec;59:99-103. doi: 10.1016/j.jsat.2015.07.002. Epub 2015 Jul 14. PMID 26254317
- [Derived] Stein MD, Anderson BJ, Thurmond P, Bailey GL. Comparing the life concerns of prescription opioid and heroin users. J Subst Abuse Treat. 2015 Jan;48(1):43-8. doi: 10.1016/j.jsat.2014.07.001. Epub 2014 Jul 11. PMID 25171955